CLINICAL TRIAL: NCT06094907
Title: An Open Label Trial of Inhaled N,N-Dimethyltryptamine in Patients With Partial Response in Depression.
Brief Title: Safety, Tolerability and Antidepressant Effects of DMT in Patients With Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Draulio Barros de Araujo, Professor, Universidade Federal do Rio Grande do Norte
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DMTPRD
Record Dates: First submitted 2023-10-10; First posted 2023-10-23 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Depressive Disorder; Depression, Unipolar
MeSH Terms: conditions — Depressive Disorder | interventions — N,N-Dimethyltryptamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- N,N-Dimethyltryptamine (Experimental): Administration of up to 2 inhaled doses of DMT within a single day (15 mg, followed by 60 mg) with a 1-hour dose interval.
  Interventions: Drug: N,N-Dimethyltryptamine

INTERVENTIONS:
Drug: N,N-Dimethyltryptamine — DMT will be administered using a vaporizer device in an ascending fixed-order of 15mg and 60mg.
  Other Names: DMT

SUMMARY:
This study aims to evaluate the acute and subacute effects of an inhaled N, N-Dimethyltryptamine (DMT) in patients with partial response in depression.

DETAILED DESCRIPTION:
This is a phase II open-label, single-ascending, fixed-order study to assess the feasibility and efficacy of inhaled N, N-Dimethyltryptamine (DMT) in patients with partial response in depression.

ELIGIBILITY:
Inclusion Criteria:

* Patients in current treatment for depression with a partial response.

Exclusion Criteria:

* heart failure
* liver failure
* kidney failure
* uncontrolled high blood pressure
* history of heart rhythm disorders
* history of valvular heart disease
* history of chronic obstructive pulmonary disease (COPD)
* active or in treatment for bronchial asthma
* severe obesity
* coagulation disorders
* clinical evidence or history of increased intracranial
* clinical evidence or history of cerebrospinal pressure
* history or reports of epilepsy
* severe neurological disease
* pregnancy
* reported or clinically recognized thyroid disorders
* diagnosis or family suspicion of genetic monoamine deficiency oxidase
* previous adverse response to psychedelic substances
* symptoms or family members with a present or past psychotic disorder
* dissociative identity disorder
* bipolar affective disorder
* prodromal symptoms of schizophrenia
* problematic use or abuse of alcohol or other psychoactive substances (except tobacco)
* acute or subacute risk of suicide
* acute flu symptoms
* symptoms of airway infection
* contact with a confirmed case of COVID-19 (SARS-CoV-2) in the last 7 days

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2023-10-09 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Change in MADRS scores | 7 days
  Change in MADRS scores from baseline to 7 days after the dosing session. The Montgomery and Asberg Depression Rating Scale (MADRS) is in portuguese and has 10 items, with an overall score ranging from 0 to 60 points. Higher score indicates more severe depression.

SECONDARY OUTCOMES:
Change in PHQ-9 scores | 7 days
  Change in PHQ-9 scores from baseline to 7 days after the dosing session. The Patient Health Questionnaire-9 (PHQ-9) is a questionnaire self-reported assessing the severity of the depression. The scale was in french and has 9 items, with an overall score ranging from 0 to 27 points. Higher score indicates more severe depression.
Change in BSI scores. | 1 day
  Change in BSI scores from baseline to 1 day after the dosing session. The Beck rating scale for suicidal ideation (BSI) is a 21-item self-report questionnaire. Each item is rated on a scale from 0 to 2, resulting in a total score ranging from 0 to 38.
Change in MADRS scores 14 days | 14 days
  Change in MADRS scores from baseline to 14 day after the dosing session. The Montgomery and Asberg Depression Rating Scale (MADRS) is in portuguese and has 10 items, with an overall score ranging from 0 to 60 points. Higher score indicates more severe depression.
Change in MADRS scores 1 month | 1 month
  Change in MADRS scores from baseline to one month after the dosing session. The Montgomery and Asberg Depression Rating Scale (MADRS) is in portuguese and has 10 items, with an overall score ranging from 0 to 60 points. Higher score indicates more severe depression.
Change in MADRS scores 3 months | 3 months
  Change in MADRS scores from baseline to three months after the dosing session. The Montgomery and Asberg Depression Rating Scale (MADRS) is in portuguese and has 10 items, with an overall score ranging from 0 to 60 points. Higher score indicates more severe depression.

OTHER OUTCOMES:
Systolic Blood Pressure | up to 2 hours
  Assessed 7 times on each session
Diastolic Blood Pressure | up to 2 hours
  Assessed 7 times on each session
Heart rate | up to 2 hours
  Assessed 7 times on each session
Respiratory rate | up to 2 hours
  Assessed 7 times on each session
Oxygen saturation | up to 2 hours
  Assessed 7 times on each session
Plasma level of C-reactive protein (CRP) | up to 2 hours
  Assessed 2 times on each session
Plasma level of cortisol | up to 2 hours
  Assessed 2 times on each session
Plasma level of brain derived neurotrophic factor | up to 2 hours
  Assessed 2 times on each session
Plasma level of glucose | up to 2 hours
  Assessed 2 times on each session
Plasma level of total cholesterol | up to 2 hours
  Assessed 2 times on each session
Plasma level of urea | up to 2 hours
  Assessed 2 times on each session
Plasma level of creatinine | up to 2 hours
  Assessed 2 times on each session
Plasma level of aspartate transaminase (AST) | up to 2 hours
  Assessed 2 times on each session
Plasma level of alanine transaminase (ALT) | up to 2 hours
  Assessed 2 times on each session
Evaluate the subjective effects of DMT | up to 2 hours
  Assessment of the acute subjective effects of DMT, by 5D-ASC (5 Dimensions - Altered States of consciousness). Scores range from 0 to 94, where higher scores indicate more intense psychedelic subjective effects.
Evaluate the mystical effects of DMT | up to 2 hours
  Assessment of the acute subjective effects of DMT, by MEQ (Questionnaire of Mystical Experiences). Scores range from 0 to 150, where higher scores indicate more intense psychedelic subjective effects.
Evaluate the influence of expectations on improvement in depressive symptoms | up to 0.5 hours
  Assessment of the influence of patient's expectations on improvement in depressive symptoms as measured by a 5 point likert scale range from: nothing to extreme.
Evaluate the influence of personality trait, by BFI (Big Five Inventory) | up to 3 months
  Assessment of the influence of personality trait assessed by the 44-item Big Five Inventory that measures an individual on the Big Five Factors (dimensions) of personality on depressive symptoms. The 5 dimensions are: Extraversion vs. introversion; Agreeableness vs. antagonism; Conscientiousness vs. lack of direction; Neuroticism vs. emotional stability; Openness vs. closedness to experience.

CONTACTS AND LOCATIONS:
Overall Officials: Draulio Araujo, Ph.D, Principal Investigator — Universidade Federal do Rio Grande do Norte; Marcelo Falchi, M.D., Study Director — Universidade Federal do Rio Grande do Norte; Fernanda Palhano-Fontes, Ph.D, Study Director — Universidade Federal do Rio Grande do Norte
Locations (1):
- Hospital Universitário Onofre Lopes, Natal, Rio Grande do Norte, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Falchi-Carvalho M, Barros H, Bolcont R, Laborde S, Wiessner I, Ruschi B Silva S, Montanini D, Barbosa DC, Teixeira E, Florence-Vilela R, Almeida R, de Macedo RKA, Arichelle F, Pantrigo EJ, Costa-Macedo JV, Arcoverde E, Galvao-Coelho N, Araujo DB, Palhano-Fontes F. The Antidepressant Effects of Vaporized N,N-Dimethyltryptamine: An Open-Label Pilot Trial in Treatment-Resistant Depression. Psychedelic Med (New Rochelle). 2025 Feb 27;3(1):48-52. doi: 10.1089/psymed.2024.0002. eCollection 2025 Mar. PMID 40337754
- [Derived] Falchi-Carvalho M, Palhano-Fontes F, Wiessner I, Barros H, Bolcont R, Laborde S, Ruschi B Silva S, Montanini D, C Barbosa D, Teixeira E, Florence-Vilela R, Almeida R, K A de Macedo R, Arichelle F, J Pantrigo E, V Costa-Macedo J, da Cruz Nunes JA, de Araujo Costa Neto LA, Nunes Ferreira LF, Dantas Correa L, da Costa Bezerra RB, Arcoverde E, Galvao-Coelho N, B Araujo D. Rapid and sustained antidepressant effects of vaporized N,N-dimethyltryptamine: a phase 2a clinical trial in treatment-resistant depression. Neuropsychopharmacology. 2025 May;50(6):895-903. doi: 10.1038/s41386-025-02091-6. Epub 2025 Apr 22. PMID 40258990